CLINICAL TRIAL: NCT03970148
Title: YAG Laser Vitreolysis of Symptomatic Vitreal Floaters
Brief Title: YAG Laser Vitreolysis for Floaters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Split (Other)
Collaborators: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Assist. prof. Ljubo Znaor, MD PhD, Principal Investigator, University Hospital of Split
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2181-147-01/06/M.S.-19-2
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Vitreous Detachment
MeSH Terms: conditions — Vitreous Detachment | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nd: YAG laser treatment (Experimental): Before treatment an optical coherence tomography (OCT) scan of the macula is performed to monitor possible macular oedema. After application of anesthetic and midriatics drops, the patient is positioned on the chin and forhead support (ND: YAG laser). Then, a contact lens (panfundoscope) is filled with methylcellulose and placed on the cornea. The laser is focused on the opacity that is to be treated and the first laser stamp of an initial power of 3 mJ is applied. The measured direct effect will guide in further adjustment of the laser beam power to achieve the desired effect. After treatment, a single drop of corticosteroid is applied to the patient and an ocular patch is applied. On follow up days an OCT scan of the macula is performed to monitor possible side effects.
  Interventions: Procedure: Nd: YAG laser

INTERVENTIONS:
Procedure: Nd: YAG laser — Before treatment an optical coherence tomography (OCT) scan of the macula is performed to monitor possible macular oedema. After application of anesthetic and midriatics drops, the patient is positioned on the chin and forhead support (ND: YAG laser). Then, a contact lens (panfundoscope) is filled with methylcellulose and placed on the cornea. The laser is focused on the opacity that is to be treated and the first laser stamp of an initial power of 3 mJ is applied. The measured direct effect will guide in further adjustment of the laser beam power to achieve the desired effect. After treatment, a single drop of corticosteroid is applied to the patient and an ocular patch is applied. On follow up days an OCT scan of the macula is performed to monitor possible side effects.

SUMMARY:
Vitreous fluid, containing 95% water, fills the space behind the lens. Its gelatinous consistency is due to the presence of hyaluronic acid, mucopolysaccharide and collagen fibers. With age, the collagen aggregates into parallel bundles, bound by cross links, leaving the pockets of liquid in the glass body. This redistribution is referred to as syneresis, which is found in 90% older than 40 years. After liquefaction, the vitreous enters the retroviral space and separates the posterior hyaloid membrane from the retina. When separating from the optical disk it forms an annular formation (Weiss ring) in front of the optical disc. These agglomerated collagen bundles (opacities) disperse the photons of light and are perceived by the patients as a "gray silhouette-like artifact". Two major interventions for these symptoms include Nd: YAG laser vitreolysis and vitrectomy. The less invasive method Nd: YAG laser increases the temperature of the opacity thus vaporizing them to smaller fragments that are easier to sediment onto the bottom of the vitreous cavity thereby relieving the symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Is able to give written informed consent to the procedure
* Patients with clinical symptoms of floaters and clinically confirmed diagnosis of opacity in the vitreous body.

Exclusion Criteria:

* Inability to tolerate the procedure
* Blurred anterior eye segment
* Cataract or Intraocular lens opacity
* Blurred posterior eye segment
* Active eye inflammation
* Iris synechiae
* Uncontrolled intraocular pressure elevation
* Peripheral retinal degeneration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-10-02 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with resolution of symptoms | 1 month
  Number of patients who reported resolution of symptoms after the treatment

SECONDARY OUTCOMES:
Macular Oedema Development rate | 1 month
  Rate of macular oedema development after the treatment
Rate of treatment side effects | 1 month
  Rate of treatment side effects such as: retinal damage, retinal detachment, cataract...
Retreatment rate | 1 month
  Number of treatment sessions needed for simptom resolution

CONTACTS AND LOCATIONS:
Overall Officials: Ljubo Znaor, MD, PHD, Principal Investigator — University Hospital of Split
Locations (1):
- University Hospital of Split, Split, Hrvatska, Croatia

IPD SHARING:
Plan to Share IPD: No